CLINICAL TRIAL: NCT06895967
Title: A Phase 1, Randomized, Open-Label, Pharmacokinetic Trial of TAK-881 and HyQvia in Healthy Adults
Brief Title: A Study of TAK-881 and HyQvia in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-881-1002
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TAK-881 1.0 g/kg (Experimental): Participants will receive TAK-881, 1.0 gram per Kilogram (g/kg), single subcutaneous (SC) injection using investigational needle sets on Day 1.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- HyQvia 1g/kg (Experimental): Participants will receive HyQvia, 1.0 g/kg, single SC injection using investigational needle sets on Day 1.
  Interventions: Biological: HyQvia; Device: SC Investigational Needle Sets

INTERVENTIONS:
Biological: TAK-881 — Participants will receive SC infusion of TAK-881.
  Other Names: Immune Globulin Subcutaneous (Human); 20% Solution with Recombinant Human Hyaluronidase (rHuPH20)
  Arms: TAK-881 1.0 g/kg
Biological: HyQvia — Participants will receive SC infusion of HyQvia.
  Other Names: Immune Globulin Subcutaneous (Human); 10% Solution with rHuPH20
  Arms: HyQvia 1g/kg
Device: SC Investigational Needle Sets — The single-use only SC needle set will be used to administer TAK-881 to the target depth below the skin surface. One needle set (single or bifurcated) will be used per infusion.
  Arms: TAK-881 1.0 g/kg
Device: SC Investigational Needle Sets — The single-use only SC needle set will be used to administer HyQvia to the target depth below the skin surface. One needle set (single or bifurcated) will be used per infusion.
  Arms: HyQvia 1g/kg

SUMMARY:
The main aim of this study is to understand how the body absorbs, processes, and removes (known as pharmacokinetics or PK) TAK-881 and HyQvia, after they are given as a single injection under the skin in healthy adults.

Study participants will receive a single dose of TAK-881 or HyQvia on Day 1.

During the study, participants will need to stay at the clinic for 8 days followed by 8 ambulatory follow up visits till Day 85.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women between 18 and 50 years can participate.
2. Must be a non-smoker, with no use of nicotine or tobacco products.
3. Must have Body Mass Index (BMI) between 18.0 and 30.0, and body weight under 120 kilograms (kg).
4. Must be medically healthy.
5. Must follow protocol-specified contraception guidance.

Exclusion Criteria:

1. Any current or past medical history of blood/clotting disorder, liver, lung, heart, kidney, immune, skin, or brain or psychiatric condition.
2. History of alcohol or drug abuse within 2 years before dosing.
3. History or presence of hypersensitivity or severe allergic reactions to blood or blood components.
4. History or presence of thrombotic/thromboembolic events, or venous thrombosis.
5. Pregnant or breastfeeding.
6. Unable to refrain from taking prescription and non-prescription medications, herbal remedies, homeopathic preparations, or vitamin supplements.
7. Recently donated blood or blood products.
8. Participated in another clinical trial involving immunoglobulin products within 12 months of screening.
9. Has taken biologic agents within 12 weeks of screening.
10. Has used an investigational product within 30 days or 5 half-lives, whichever is longer, prior to screening.
11. Has received any vaccine (including live attenuated vaccines and COVID-19 vaccines) during the last 30 days before dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Baseline-corrected Area Under the Concentration-time Curve (AUC) From Day 1 to Day 29 (AUC Day1-29) Based on Serum Total Immunoglobulin G (IgG) Levels | Day 1 up to Day 29

SECONDARY OUTCOMES:
Baseline-Uncorrected Maximum Observed Concentration (Cmax) Based on Serum Total IgG Levels | From Screening up to Day 85
Baseline-Uncorrected Time to Maximum Concentration (Tmax) Based on Serum Total IgG Levels | From Screening up to Day 85
Baseline-Uncorrected AUC Day1-29 Based on Serum Total IgG Levels | Day 1 up to Day 29
Baseline-corrected AUC from Day 1 to infinity (AUCinf) Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected AUC from Day 1 to Time of the Last Measurable Concentration (AUClast) Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Cmax Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Tmax Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Time of last measurable concentration (Tlast) Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Terminal Half-life (t1/2z) Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Apparent Clearance (CL/F) Based on Serum Total IgG Levels | From Day 1 up to Day 85
Baseline-corrected Apparent Volume of Distribution (Vz/F) Based on Serum Total IgG Levels | From Day up to Day 85
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug up to Day 85
  TEAEs are defined as AEs that started at or after the initiation of the first administration of TAK-881 or HyQvia or any adverse event already present that worsens in either intensity or frequency following exposure to TAK-881 or HyQvia.
Number of Participants With Infusion Withdrawals, Interruptions, and Infusion Rate Reductions | From first dose of study drug up to Day 85
Number of Participants With Positive Binding Antibodies to rHuPH20 | From first dose of study drug up to Day 85
Number of Participants With Neutralizing Antibodies to rHuPH20 | From first dose of study drug up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/69ac38d2f24d46be